CLINICAL TRIAL: NCT01299116
Title: Long-Acting Reversible Contraception: New Research to Reduce Unintended Pregnancy
Brief Title: Long-Acting Reversible Contraception
Acronym: LARC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: FHI 360 (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 10250
Record Dates: First submitted 2011-02-16; First posted 2011-02-18 (Estimated); Results first posted 2018-01-26 (Actual); Last update posted 2018-02-28 (Actual); Status verified 2018-01

CONDITIONS: Contraception
Keywords: AE-adverse event; FDA-(U.S.) Food and Drug Administration; GCP-Good Clinical Practice guidelines; ICH-International Committee on Harmonisation; IRB-Institutional Review Board; IU-International units; mg-milligram(s); mm3-cubic millimeter(s); LARC-Long-Acting reversible contraception; PPCNC-Planned Parenthood of North Carolina; SAE-serious adverse event; SARC-Short-Acting reversible contraception; µg-microgram; ULN-upper limit of the normal range; SubQ-subcutaneous
MeSH Terms: interventions — N,N-dimethyl-4-anisidine; Contraceptives, Oral; etonogestrel; Levonorgestrel

STUDY DESIGN:
Intervention Model Description: Partially randomized patient preference trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Preference SARC (Other): Participants received one of a variety of oral contraceptives or DMPA
  Interventions: Drug: DMPA; Drug: oral contraceptives
- Randomized LARC (Experimental): Participants receive one of the following interventions:
  Implanon® or Nexplanon®; ParaGard®; Mirena®
  Interventions: Drug: Implanon®; Drug: ParaGard®; Drug: Mirena®
- Randomized SARC (Active Comparator): Participants received one of a variety of oral contraceptives or DMPA
  Interventions: Drug: DMPA; Drug: oral contraceptives

INTERVENTIONS:
Drug: DMPA — Injectable contraceptive, containing 150 mg depot medroxyprogesterone acetate (DMPA) and marketed in the US as Depo-Provera® or containing 104 mg DMPA and marketed as Depo-SubQ Provera 104®.
  Arms: Preference SARC; Randomized SARC
Drug: oral contraceptives — Oral contraceptives (any variety of formulations are permitted)
  Arms: Preference SARC; Randomized SARC
Drug: Implanon® — Subdermal contraceptive implant, marketed in the US as Implanon® or Nexplanon® (containing 68 mg of etonogestrel)
  Other Names: Nexplanon®
  Arms: Randomized LARC
Drug: ParaGard® — Intrauterine device marketed in the US as ParaGard® (a T-shaped plastic device containing 380mm2 of copper surface)
  Arms: Randomized LARC
Drug: Mirena® — Intrauterine system, marketed in the US as Mirena® (containing 52 mg of levonorgestrel)
  Arms: Randomized LARC

SUMMARY:
In the proposed study, women aged 18-29 seeking oral or injectable contraception will be offered an opportunity to try LARC instead; the FDA-approved options include two types of intrauterine products and one type of subdermal contraceptive implant. Over a 24 month period, the experiences of LARC users will be compared to the experiences of those opting for their initial short-acting method.

DETAILED DESCRIPTION:
In this partially randomized patient preference study, women aged 18-29 seeking oral or injectable contraception will be offered an opportunity to try LARC instead; the FDA-approved options include two types of intrauterine products and one type of subdermal contraceptive implant. Over a 24-month period, the experiences of LARC users will be compared to the experiences of those opting for their initial short-acting method. It is expected that 38% of the participants using short-acting methods will stop using them during the first year and be at risk of unintended pregnancy. In contrast, less than 20% of LARC users will want to have their contraceptive removed. Continuation rates will be measured and pregnancies will be tallied in the two groups to document any differences that emerge.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 29 years of age;
* sexually active;
* seeking oral or injectable contraception;
* working cell phone;
* working email account;
* willingness to be contacted by the clinic staff or study coordinators; and,
* willingness to complete questionnaires.

Exclusion Criteria:

* currently pregnant;
* previous use of a long-acting reversible contraceptive (LARC) method; and,
* medical contraindications for oral contraceptives and injectables.

Ages: 18 Years to 29 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 916 (Actual)
Dates: Start 2011-12 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Hubacher, PhD, Principal Investigator — FHI 360
Locations (1):
- Planned Parenthood Central North Carolina, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hubacher D, Spector H, Monteith C, Chen PL, Hart C. Long-acting reversible contraceptive acceptability and unintended pregnancy among women presenting for short-acting methods: a randomized patient preference trial. Am J Obstet Gynecol. 2017 Feb;216(2):101-109. doi: 10.1016/j.ajog.2016.08.033. Epub 2016 Sep 20. PMID 27662799
- [Background] Hubacher D, Spector H, Monteith C, Chen PL, Hart C. Rationale and enrollment results for a partially randomized patient preference trial to compare continuation rates of short-acting and long-acting reversible contraception. Contraception. 2015 Mar;91(3):185-92. doi: 10.1016/j.contraception.2014.11.006. Epub 2014 Nov 15. PMID 25500324
- [Derived] Burke HM, Packer CA, Spector HL, Hubacher D. Opportunity, satisfaction, and regret: Trying long-acting reversible contraception in a unique scientific circumstance. Women Health. 2019 Mar;59(3):266-280. doi: 10.1080/03630242.2018.1478363. Epub 2018 Aug 1. PMID 29920171
- [Derived] Hubacher D, Spector H, Monteith C, Chen PL. Not seeking yet trying long-acting reversible contraception: a 24-month randomized trial on continuation, unintended pregnancy and satisfaction. Contraception. 2018 Jun;97(6):524-532. doi: 10.1016/j.contraception.2018.02.001. Epub 2018 Feb 19. PMID 29470950

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is a partially randomized patient preference trial. Twenty two participants did not contribute data for analysis because they did not start a contraceptive in one of the three groups. For more information see: Hubacher D et al., 2017. The total number going forward for analysis is 894.
Groups:
- SARC - Preference: Participants received one of a variety of oral contraceptives or DMPA
  DMPA: Injectable contraceptive, containing 150 mg depot medroxyprogesterone acetate (DMPA) and marketed in the US as Depo-Provera® or containing 104 mg DMPA and marketed as Depo-SubQ Provera 104®.
  oral contraceptives: Oral contraceptives (any variety of formulations are permitted)
- LARC - Randomized: Participants receive one of the following interventions:
  Implanon® or Nexplanon®; ParaGard®; Mirena®
  Implanon®: Subdermal contraceptive implant, marketed in the US as Implanon® or Nexplanon® (containing 68 mg of etonogestrel)
  ParaGard®: Intrauterine device marketed in the US as ParaGard® (a T-shaped plastic device containing 380mm2 of copper surface)
  Mirena®: Intrauterine system, marketed in the US as Mirena® (containing 52 mg of levonorgestrel)
- SARC - Randomized: Participants received one of a variety of oral contraceptives or DMPA
  DMPA: Injectable contraceptive, containing 150 mg depot medroxyprogesterone acetate (DMPA) and marketed in the US as Depo-Provera® or containing 104 mg DMPA and marketed as Depo-SubQ Provera 104®.
Period: Overall Study
Arm/Group | SARC - Preference | LARC - Randomized | SARC - Randomized
Started | 522 | 177 | 195
Completed | 457 | 168 | 184
Not Completed | 65 | 9 | 11
Not completed — Lost to Follow-up | 65 | 9 | 11

BASELINE CHARACTERISTICS:
Groups:
- Randomized LARC: Participants receive one of the following interventions:
  Implanon® or Nexplanon®; ParaGard®; Mirena®
  Implanon®: Subdermal contraceptive implant, marketed in the US as Implanon® or Nexplanon® (containing 68 mg of etonogestrel)
  ParaGard®: Intrauterine device marketed in the US as ParaGard® (a T-shaped plastic device containing 380mm2 of copper surface)
  Mirena®: Intrauterine system, marketed in the US as Mirena® (containing 52 mg of levonorgestrel)
- Total: Total of all reporting groups
Arm/Group | Preference SARC | Randomized LARC | Randomized SARC | Total
Number analyzed (Participants) | 522 | 177 | 195 | 894
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 23 [21 to 26] | 23 [21 to 26] | 23 [21 to 26] | 23 [21 to 26]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 522 | 177 | 195 | 894
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Three participants did not provide race/ethnicity information
  Participants
    Hispanic | 68 | 14 | 30 | 112
    Non-Hispanic, white | 269 | 111 | 105 | 485
    Non-Hispanic, black | 124 | 34 | 44 | 202
    All other single and multiple race | 58 | 18 | 16 | 92

OUTCOME MEASURES:

1. Primary Outcome: Contraceptive Method Discontinuation
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | SARC - Preference | LARC - Randomized | SARC - Randomized
Number analyzed (Participants) | 522 | 177 | 195
Participants | 300 | 62 | 142

2. Secondary Outcome: Unintended Pregnancy
Description: Intent-to-treat principles applied.
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | SARC - Preference | LARC - Randomized | SARC - Randomized
Number analyzed (Participants) | 466 | 168 | 187
Participants | 47 | 6 | 13

3. Secondary Outcome: Participant Attitudes to LARC vs SARC
Description: Level of happiness with initial method (% distribution)
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Preference SARC | Randomized LARC | Randomized SARC
Number analyzed (Participants) | 522 | 177 | 195
Participants
  Happy | 354 | 120 | 138
  Neutral | 52 | 15 | 24
  Unhappy | 50 | 33 | 22
  Missing | 66 | 9 | 11

ADVERSE EVENTS:
Time Frame: 24 months
Description: Only serious adverse events were collected. AEs not captured.
Arm/Group | SARC - Preference | LARC - Randomized | SARC - Randomized
All-Cause Mortality (participants affected / at risk) | 0/522 | 0/177 | 0/195
Serious Adverse Events (participants affected / at risk) | 0/522 | 1/177 | 0/195
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SARC - Preference (N=522) | LARC - Randomized (N=177) | SARC - Randomized (N=195)
endometritis (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes